CLINICAL TRIAL: NCT03502928
Title: Efficacy of the Use of Dry Needling in Conventional Non-invasive Treatment of Acute and Subacute Whiplash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Raquel Lorenzo Moreno, physiotherapist, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1489327794181094
Record Dates: First submitted 2018-04-05; First posted 2018-04-19 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Whiplash Injuries
Keywords: Dry Needling; Manual Therapy; Motor Control; Whiplash
MeSH Terms: conditions — Whiplash Injuries | interventions — Functional Laterality; Musculoskeletal Manipulations; Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (Active Comparator): Motor Control + Manual Therapy
  Interventions: Other: Motor Control; Other: Manual Therapy
- Experimental Treatment (Experimental): Motor Control + Manual Therapy + Dry Needling
  Interventions: Other: Motor Control; Other: Manual Therapy; Other: Dry Needling

INTERVENTIONS:
Other: Motor Control — Neck Motor Control
Other: Manual Therapy — Massage + Joint Mobilizations
Other: Dry Needling — Dry Needling in Neck Muscles
  Arms: Experimental Treatment

SUMMARY:
INTRODUCTION: Whiplash is an injury produced by an acceleration-deceleration mechanism that transmits energy to the cervical spine. According to the bibliography, the conservative treatment (motor control exercises and manual therapy) has shown benefits in approaching this lesion, but its efficacy is limited. Dry needling has already shown its usefulness in different musculoskeletal pathologies, however, its efficacy is unknown when it is included in conservative treatment.

OBJECTIVES: The objective of this study is to assess the effects of the incorporation of dry needling in the conventional treatment with manual therapy and motor control exercises, compared to the conventional non-invasive treatment in patients with acute or subacute whiplash.

HYPOTHESIS: The inclusion of dry needling in conventional non-invasive treatment is more effective than conventional non-invasive treatment in patients with acute or subacute whiplash.

METHODS: A randomized clinical trial will be conducted in which the subjects of study will be assigned to two groups, a control group (conventional treatment) and an experimental group (conventional treatment and dry needling).

ELIGIBILITY:
Inclusion Criteria:

* Medical Diagnosis of Whiplash Grade I-II in the QTF
* Neck Pain
* Whiplash in Acute or Subacute Phase

Exclusion Criteria:

* Pregnancy
* Belonephobia
* Cervical Fractures-Dislocations or Neurological Deficit Secondaries to Accident
* Previous Surgery of the Cervical Spine
* Circulatory Disease, Respiratory Disease, Neurological Disease, Rheumatologic Disease and Mental Illness
* Athletes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index. Changes from Baseline | 3 weeks, 6 weeks, 3 months
  0-100% (0% = No Disability; 100% = Disability (highest level of disability)

SECONDARY OUTCOMES:
Pressure pain thresholds. Changes from Baseline | 3 weeks, 6 weeks, 3 months
  The minimum force applied which induces pain. Measured kg/cm2
Cervical Range of Movement. Changes from Baseline | 3 weeks, 6 weeks, 3 months
  Amount of cervical movement using a goniometer
Kinesophobia. Changes from Baseline | 3 weeks, 6 weeks, 3 months
  Fear of movement measured by the TAMPA scale
Cervical Motor Control. Changes from Baseline | 3 weeks, 6 weeks, 3 months
  measure of cervical joint position sense using a laser

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Achalandabaso, PhD, Study Director — University of Jaén
Locations (1):
- Universidad de Alcalá, Alcalá de Henares, Spain

IPD SHARING:
Plan to Share IPD: No